CLINICAL TRIAL: NCT02037724
Title: Fermented Iron-rich Supplement in Reducing Anemia
Acronym: FISRA
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Ghana (Other)
Responsible Party: Principal Investigator, Richmond Aryeetey, PhD, MPH, Senior Lecturer, University of Ghana
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UG-0001-IDA
Record Dates: First submitted 2014-01-14; First posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2014-01

CONDITIONS: Iron Deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Iron-Dextran Complex; Iron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- supplement containing 60 mg iron sulfate (Other): nutrient supplement containing 60 mg of iron as ferous sulfate
  Interventions: Dietary Supplement: iron rich food supplement (60 mg iron); Dietary Supplement: iron rich food supplement (10 mg iron); Dietary Supplement: supplement containing 10 mg iron sulfate
- iron rich food supplement (60 mg iron) (Experimental): contains 60 mg Iron
  Interventions: Dietary Supplement: supplement containing 60 mg iron sulfate; Dietary Supplement: iron rich food supplement (10 mg iron); Dietary Supplement: supplement containing 10 mg iron sulfate
- iron rich food supplement (10 mg iron) (Experimental): contains 10 mg of iron
  Interventions: Dietary Supplement: supplement containing 60 mg iron sulfate; Dietary Supplement: iron rich food supplement (60 mg iron); Dietary Supplement: supplement containing 10 mg iron sulfate
- supplement containing 10 mg iron sulfate (Other): nutrient supplement containing 10 mg of iron as ferous sulfate
  Interventions: Dietary Supplement: supplement containing 60 mg iron sulfate; Dietary Supplement: iron rich food supplement (60 mg iron); Dietary Supplement: iron rich food supplement (10 mg iron)

INTERVENTIONS:
Dietary Supplement: supplement containing 60 mg iron sulfate — control agent
  Arms: iron rich food supplement (10 mg iron); iron rich food supplement (60 mg iron); supplement containing 10 mg iron sulfate
Dietary Supplement: iron rich food supplement (60 mg iron) — contains 60 mg of iron
  Arms: iron rich food supplement (10 mg iron); supplement containing 10 mg iron sulfate; supplement containing 60 mg iron sulfate
Dietary Supplement: iron rich food supplement (10 mg iron) — contains 10 mg iron
  Arms: iron rich food supplement (60 mg iron); supplement containing 10 mg iron sulfate; supplement containing 60 mg iron sulfate
Dietary Supplement: supplement containing 10 mg iron sulfate — control agent
  Arms: iron rich food supplement (10 mg iron); iron rich food supplement (60 mg iron); supplement containing 60 mg iron sulfate

SUMMARY:
The consequences of iron deficiency anemia in women are enormous, and especially in developing countries, as the condition adversely affects both their productive and reproductive capabilities. The study seeks to: 1) compare changes in iron status indicators among women receiving an iron-rich organic food supplement versus ferrous sulfate supplement, and 2) determine the suitable level of food supplement needed to prevent/reduce iron deficiency anemia among women in developing country settings.

A double-blind, randomized, controlled, intervention trial will be implemented in women of childbearing age, 60 women with iron deficiency anemia and 60 women with iron deficiency. After screening potential subjects (up to 500 expected), approximately 30 will be recruited into each of four study groups; assuming 30% dropout rate, to detect an increase of 30% in ferritin as significant between the two time points at 80% power and alpha value of 0.05. Subjects who meet the inclusion criteria will be randomized into the four groups consisting of: 2 control groups (daily 60mg ferrous sulfate (FS-60) or daily 10mg ferrous sulfate (FS-10)), and 2 test groups (daily 60mg iron-rich supplement (IRS-60) or 10mg iron-rich supplement (IRS-10)). Subjects will take daily FS-60 and IRS-60 under supervision for 8 weeks while subjects taking FS-10 and IRS-10 will take the supplement under supervision for 12 consecutive weeks.

DETAILED DESCRIPTION:
The design will involve screening of about 500 female adult students and staff of the University of Ghana who meet initial the inclusion criteria. Screening will involve pregnancy testing, assessment of hemoglobin, and ferritin and also administration of a health history questionnaire.

Thereafter, 120 eligible subjects will enrolled and randomized to recieve the treatment. All subjects will complete 3-day dietary record (including 2 weekdays and 1 weekend) at baseline and at endline (i.e. one week prior to treatment completion). The dietary data will be analyzed using nationally-generated food composition tables together with the ESHA food processor software. In addition, body weight and height will be measured using standard methods at baseline and end of the study. Weekly monitoring of side effects will be recorded. Fasting blood samples will be collected at baseline and endline to enable determination of anemia status and other indicators including serum ferritin, transferrin receptor and full blood count, together with C-reactive protein.

ELIGIBILITY:
Inclusion Criteria:

* 18-49 years
* Regular menstruation in the last three months
* Hemoglobin <12 mg/dl;
* Serum Ferittin<20mcg/L
* BMI 18.5Kg/m^2 to 29.9 kg/m^2

Exclusion Criteria:

* history of gastrointestinal or hematological disorders,
* taking medications that could interfere with hematopoiesis or dietary iron absorption
* pregnant (based on pregnancy test).

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-08 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
iron deficiency anemia | two and three months
  Improvement of iron status with 60 mg (after two months) and 10 mg iron (after 3 months) will be assessed. The iron status measurements include, hemoglobin, ferritin, transferrin receptor and whole blood count

SECONDARY OUTCOMES:
comparison of side effects of iron supplement | 3 months
  We expect to have less side effects with IRS compared with ferrous sulfate (as observed in previous studies) that include: constipation, diarrhea, vomiting, gastrointestinal distress, change in stool color and others. We will assess these with a questionnaire.

OTHER OUTCOMES:
minimum level of supplement intake needed to improve iron status | 3 months
  The effectiveness of low dose (10 mg daily iron) compared to higher dose (60mg daily iron) from the fermented organic food supplement product. These results will be helpful for using IRS as a food supplement.

CONTACTS AND LOCATIONS:
Overall Officials: Richmond Aryeetey, PhD, Principal Investigator — University of Ghana; Manju Reddy, PhD, Principal Investigator — Iowa State University